CLINICAL TRIAL: NCT05011786
Title: Is the Open Approach Superior to the Laparoscopic Hernia Repair in Children? A Retrospective Comparative Study.
Brief Title: Open and Laparoscopic Hernia Repair. A Comparative Study
Status: Completed | Type: Observational
Sponsor: Ibrahim Khrais (Other)
Responsible Party: Sponsor-Investigator, Ibrahim Khrais, Co-investigator, University of Jordan
Organization: University of Jordan (Other)
Other Study IDs: 67-2019-5771
Record Dates: First submitted 2021-07-20; First posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-07

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal | interventions — Herniorrhaphy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Open repair group: children with inguinal hernia who were repaired with open high ligation of the hernia sac through an inguinal incision.
  Interventions: Procedure: hernia repair/ligation of the hernial sac
- Laparoscopic repair group: children with inguinal hernia who were repaired laparoscopically by closing the the PPV at the level of internal ring with a purse string suture
  Interventions: Procedure: hernia repair/ligation of the hernial sac

INTERVENTIONS:
Procedure: hernia repair/ligation of the hernial sac — the inguinal hernia sac is ligated using sutures at the level of internal ring throught an inguinal incision in the open group and using laparoscopic instruments in the laparoscopic group

SUMMARY:
A retrospective comparative study in a pediatric surgery center to compare the outcomes of 2 approaches of hernia repair in the pediatric population.

DETAILED DESCRIPTION:
The investigators reviewed the records of all children who underwent open or laparoscopic hernia repair between January 2017 and July 2019 at the pediatric surgery center at the Jordan University Hospital. Data collection included the age, gender, laterality of the hernia, the surgical approach, duration of surgery, time to discharge and time to full recovery.

ELIGIBILITY:
Inclusion Criteria:

* All children within the age limit specified were included in the study

Exclusion Criteria:

* none

Ages: 6 Months to 13 Years | Sex: All
Age Groups: Child
Study Population: all children aged between 6 months and 13 years who underwent open or laparoscopic inguinal hernia repair at the Jordan University Hospital in the period between January 2017 and July 2019
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
OR duration | During surgery
Length of stay LOS | 1 year
Post operative complications | 1 year
Hernia Recurrence | 1 year
Total Cost of Surgery | 1 year
Cosmesis | 1 Year
  What does the parents of the children think of the cosmetic outcomes of the surgery on a scale from 1-5
Recovery | year
  Time from discharge to resuming normal daily activities

CONTACTS AND LOCATIONS:
Locations (1):
- Ibrahim Khrais, Amman, Please Select, Jordan

IPD SHARING:
Plan to Share IPD: Undecided